CLINICAL TRIAL: NCT03891654
Title: Pilot Study of Dynamic Contrast Enhanced Computed Tomography (DCE-CT) Imaging for the Assessment of Radiation Therapy Outcome for Liver Cancer Patients
Brief Title: Dynamic Contrast Enhanced Computed Tomography to Assess Radiation Therapy in Liver Cancer Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-2874.cc; P30CA046934 (NIH)
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Liver Cancer
Keywords: Radiation; Metastases; Dynamic Contrast Enhanced Computed Tomography; Pilot
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Each patient will receive the standard of care, with the intervention, DCE-CT perfusion, occurring pre-treatment and post-treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Dynamic Contrast Enhanced Computed Tomography (Experimental): DCE-CT, also known as perfusion CT, is a functional imaging modality that uses repeated computed tomography imaging after injection of an iodine based contrast agent.
  Interventions: Diagnostic Test: Dynamic Contrast Enhanced Computed Tomography

INTERVENTIONS:
Diagnostic Test: Dynamic Contrast Enhanced Computed Tomography — Patients will receive DCE-CT prior to the start of standard of care, Stereotactic Body Radiation Therapy (SBRT), as well as 6 hours post administration of SBRT and 6 weeks post administration of SBRT.
  Other Names: DCE-CT; Perfusion CT

SUMMARY:
This is a pilot study that uses a standard of care technique, Stereotactic Body Radiation Therapy (SBRT), in combination with Dynamic Contrast Enhanced Computed Tomography (DCE-CT) to determine if perfusion changes from SBRT of liver cancer may be used for outcome assessment and prediction of prognosis.

DETAILED DESCRIPTION:
Patients will undergo standard of care SBRT while also receiving DCE-CT, also known as perfusion CT, pre-treatment, 6 hours post-treatment and 6 weeks post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form
2. Stated willingness to comply with all study procedures and be available for the duration of the study
3. Be a Male or Female aged 18-100
4. Diagnosed with Liver HCC or metastases
5. Must be receiving or will plan to receive SBRT for Liver HCC or metastases

Exclusion Criteria:

1. Allergy to iodine contrast
2. CT with contrast not offered as a Standard of Care
3. Pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
DCE-CT Perfusion Metrics: K-Trans | Baseline to end of follow-up, up to 12 weeks
  Determine the association between the delivered radiation therapy dose distribution and the change in perfusion measurement through K-Trans (extraction-flow product) as shown through DCE-CT imaging.
DCE-CT Perfusion Metrics: Blood Volume | Baseline to end of follow-up, up to 12 weeks
  Determine the association between the delivered radiation therapy dose distribution and the change in perfusion measurement through blood volume as shown through DCE-CT imaging.
DCE-CT Perfusion Metrics: Blood Flow | Baseline to end of follow-up, up to 12 weeks
  Determine the association between the delivered radiation therapy dose distribution and the change in perfusion measurement through blood flow as shown through DCE-CT imaging.

SECONDARY OUTCOMES:
Correlation Between Patient Demographics and K-Trans: Age | Post follow-up to end of study, up to 12 months
  Stratify K-Trans results by age to determine correlation of DCE-CT imaging results compared to patient demographics
Correlation Between Patient Demographics and K-Trans: Sex | Post follow-up to end of study, up to 12 months
  Stratify K-Trans results by sex to determine correlation of DCE-CT imaging results compared to patient demographics
Correlation Between Patient Demographics and K-Trans: Race | Post follow-up to end of study, up to 12 months
  Stratify K-Trans results by race to determine correlation of DCE-CT imaging results compared to patient demographics
Correlation Between Patient Demographics and K-Trans: Clinical Stage of Disease | Post follow-up to end of study, up to 12 months
  Stratify K-Trans results by clinical stage at diagnosis to determine correlation of DCE-CT imaging results compared to patient demographics
Correlation Between Patient Demographics and Blood Volume: Age | Post follow-up to end of study, up to 12 months
  Stratify blood volume results age to determine correlation of DCE-CT imaging results compared to patient demographics
Correlation Between Patient Demographics and Blood Volume: Sex | Post follow-up to end of study, up to 12 months
  Stratify blood volume results sex to determine correlation of DCE-CT imaging results compared to patient demographics
Correlation Between Patient Demographics and Blood Volume: Race | Post follow-up to end of study, up to 12 months
  Stratify blood volume results race to determine correlation of DCE-CT imaging results compared to patient demographics
Correlation Between Patient Demographics and Blood Volume: Clinical Stage of Disease | Post follow-up to end of study, up to 12 months
  Stratify blood volume results by clinical stage at diagnosis to determine correlation of DCE-CT imaging results compared to patient demographics
Correlation Between Patient Demographics and Blood Flow: Age | Post follow-up to end of study, up to 12 months
  Stratify blood flow results age to determine correlation of DCE-CT imaging results compared to patient demographics
Correlation Between Patient Demographics and Blood Flow: Sex | Post follow-up to end of study, up to 12 months
  Stratify blood flow results sex to determine correlation of DCE-CT imaging results compared to patient demographics
Correlation Between Patient Demographics and Blood Flow: Race | Post follow-up to end of study, up to 12 months
  Stratify blood flow results race to determine correlation of DCE-CT imaging results compared to patient demographics
Correlation Between Patient Demographics and Blood Flow: Clinical Stage of Disease | Post follow-up to end of study, up to 12 months
  Stratify blood flow results by clinical stage at diagnosis to determine correlation of DCE-CT imaging results compared to patient demographics

CONTACTS AND LOCATIONS:
Overall Officials: Moyed Miften, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT03891654/Prot_SAP_ICF_000.pdf